CLINICAL TRIAL: NCT04535895
Title: Simultaneous Integrated Boost (SIB) Technique in the Adjuvant Radiotherapy of Breast Cancer Patients.
Brief Title: Simultaneous Integrated Boost Technique in Breast Cancer Radiotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Treatment standard has changed
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1094/2020
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous integrated boost arm (Experimental)
  Interventions: Radiation: Simultaneous integrated boost

INTERVENTIONS:
Radiation: Simultaneous integrated boost — Adjuvant breast cancer irradiation including simultaneous integrated boost

SUMMARY:
Adjuvant radiotherapy after breast conserving surgery has been shown to improve both local control and overall survival. Dose escalation of the tumor bed by addition of a boost after whole breast radiotherapy reduces the risk of local recurrence in invasive breast cancer.

Simultaneous integrated boost (SIB) techniques have been shown to provide more conformal treatment plans than conventional sequential boost, in addition, SIB enables a reduction in the overall treatment time by 1 week compared to conventional boost techniques.

The proposed study is aimed at evaluating radiation-induced toxicity in patients treated with breast-conserving surgery in combination with radiotherapy using SIB technique.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer or ductal carcinoma in situ
* Breast conserving surgery
* Complete tumor resection
* Treatment with adjuvant radiotherapy of the breast
* Indication for boost Irradiation
* Given informed consent

Exclusion Criteria:

* Incomplete tumor resection
* Mastectomy
* Distant metastases at diagnosis
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Acute Radiation induced toxicity (grade 2 or higher) | Measurement at the last 1 day of radiotherapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Acute Radiation induced toxicity (grade 2 or higher) | Measurement 3 months after completion of radiotherapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Langsenlehner, MD, Principal Investigator — Medical University of Graz, Dept. of Therapeutic Radiology and Oncology
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurkmans CW, Dijckmans I, Reijnen M, van der Leer J, van Vliet-Vroegindeweij C, van der Sangen M. Adaptive radiation therapy for breast IMRT-simultaneously integrated boost: three-year clinical experience. Radiother Oncol. 2012 May;103(2):183-7. doi: 10.1016/j.radonc.2011.12.014. Epub 2012 Jan 24. PMID 22280808